CLINICAL TRIAL: NCT05372250
Title: Assessment of the Impact of Body Position on Diaphragmatic Excursion in Obese Patients to Improve Proactice in Respiratory Kinesitherapy
Acronym: EXDECHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Marine MERVELET, Principal Investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A00063-40
Record Dates: First submitted 2022-04-27; First posted 2022-05-12 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Order of body positions for ultrasound measurements : supine position, 45°, sitting, standing (Experimental)
  Interventions: Other: Measurement of the diaphragmatic excursion according to the position of the body by ultrasound
- Order of body positions for ultrasound measurements : 45°, sitting, standing, supine position. (Experimental)
  Interventions: Other: Measurement of the diaphragmatic excursion according to the position of the body by ultrasound
- Order of body positions for ultrasound measurements : sitting, standing, supine, 45°. (Experimental)
  Interventions: Other: Measurement of the diaphragmatic excursion according to the position of the body by ultrasound
- Order of body positions for ultrasound measurements : standing, supine, 45°, seated. (Experimental)
  Interventions: Other: Measurement of the diaphragmatic excursion according to the position of the body by ultrasound

INTERVENTIONS:
Other: Measurement of the diaphragmatic excursion according to the position of the body by ultrasound — Measurement of the diaphragmatic excursion according to the position of the body by ultrasound

SUMMARY:
The EXDECHO study is the first randomized study evaluating the effect of four body positions on diaphragmatic excursion in obese patients by ultrasound.

The investigators suppose that the course of the right diaphragmatic hemicupola would be increased by an increasingly horizontal position (gradual increase in the diaphragmatic excursion from standing to lying down).

If this hypothesis is confirmed, kinesitherapists will have more informed positioning choices to improve the effectiveness of respiratory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* to have a BMI greater than or equal to 30;
* to have not had intense physical activity during the hour preceding the measurements;
* to be enrolled in a social security plan;
* to give a written consent;
* to have underwent a pre-inclusion medicalexamination.

Exclusion Criteria:

* to have a respiratory pathology unrelated to obesity (sleep apnea syndrome, obesity-hypoventilation syndrome, restrictive ventilatory syndrome with no other known cause);
* to have a cardiac pathology not stabilized by drug treatment and/or resulting in heart failure and/or requiring the fitting of a pacemaker or defibrillator;
* to have a chronic inflammatory disease (rheumatoid arthritis, Crohn's disease, cirrhosis, etc.);
* to have a chest deformity (kyphoscoliosis, funnel chest, etc.);
* to be anactive smoking or former smoker (stopped for less than 3 months and total consumption > 10 pack-years);
* to have an history of major surgery, surgery under general anesthesia for less than 3 months, or minimally invasive surgery for less than 1 year of the thoraco-abdomino-pelvic compartments;
* to have a known sensitivity to monopropylene glycol (substance present in the sterile ultrasound gel);
* temperature of the room in which the ultrasound measurements are carried out below 20°C or above 25°C;
* subject under a measure of legal protection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic excursion in centimeters in the 4 positions measured by ultrasound | Day 0

SECONDARY OUTCOMES:
Correlation between measurement of diaphragmatic excursion in centimeters by ultrasound and weight in kilograms. | Day 0
Correlation between measurement of diaphragmatic excursion in centimeters by ultrasound and waist circumference in centimeters. | Day 0
Correlation between measurement of diaphragmatic excursion in centimeters by ultrasound and BMI in kg/m². Weight in kilograms and height in meters will be combined to report BMI in kg/m². | Day 0
Correlation between measurement of diaphragmatic excursion in centimeters by ultrasound and sex of the participant (male/female). | Day 0
Comfort of the ultrasound examination felt by the patient via a questionnaire | Day 0
  Positions, duration of the examination, pressure exerted by the probe: score from 0 (unpleasant) to 4 (acceptable)

CONTACTS AND LOCATIONS:
Overall Officials: Marine Mervelet, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Vandœuvre-lès-Nancy, France